CLINICAL TRIAL: NCT07324317
Title: A Prospective Clinical Validation Study of an End-to-End Difficult Airway Pathway Planning Algorithm (EAP-LC) in Patients With Laryngeal Cancer: A Spatial Consistency Assessment Based on Awake Flexible Bronchoscopic Intubation Videos
Brief Title: Validation of End-to-End Difficult Airway Pathway Planning Algorithm (EAP-LC)
Status: Not yet recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025321
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Laryngeal Cancer; Difficult Airway
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Awake Flexible Bronchoscopic Intubation Group
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Intervention

SUMMARY:
Patients with laryngeal cancer often present with varying degrees of airway narrowing or anatomical distortion, making airway management particularly challenging. Awake flexible bronchoscopic intubation is a widely accepted and important strategy to ensure airway safety in this population. Currently, the selection of the intubation pathway mainly relies on visual assessment of preoperative computed tomography (CT) images and the clinical experience of anesthesiologists, lacking objective and quantifiable tools for airway pathway planning.

Our research group has developed an end-to-end airway pathway planning algorithm for laryngeal cancer patients (EAP-LC), which can automatically generate predicted nasal or oral intubation pathways based on preoperative pharyngeal and upper airway CT images. Preliminary simulation analyses based on retrospective CT data demonstrated that the algorithm is capable of identifying airway narrowing and generating trajectories that are close to clinically feasible intubation paths (preliminary data, under review). However, to date, no study has directly compared the algorithm-predicted pathways with actual intubation trajectories obtained during awake flexible bronchoscopic intubation. Therefore, a prospective clinical validation study is required to evaluate the spatial consistency and clinical feasibility of the EAP-LC algorithm.

Without altering routine clinical treatment or anesthetic management, this study aims to evaluate the clinical accuracy, safety, and feasibility of the EAP-LC algorithm by comparing the intubation pathways predicted from preoperative CT images with the real-world trajectories recorded during awake flexible bronchoscopic intubation. The results of this study are expected to provide a more precise and objective decision-support tool for airway management in patients with laryngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo laryngeal cancer surgery under general anesthesia, including supraglottic, glottic, and subglottic laryngeal cancers, as well as lesions involving the hypopharynx-larynx junction, who are assessed preoperatively as requiring awake flexible bronchoscopic intubation. Eligible participants must meet all of the following criteria: age ≥ 18 years, with no restriction on sex; a confirmed diagnosis of laryngeal cancer or laryngeal tumor based on previous or preoperative imaging and/or pathological findings; a planned laryngeal surgical procedure; a preoperative anesthetic assessment indicating the need for awake flexible bronchoscopic intubation to ensure airway safety; completion of contrast-enhanced laryngeal and/or cervical computed tomography (CT) within 2 weeks prior to surgery, with image quality adequate for analysis by the EAP-LC algorithm; clear consciousness, the ability to understand the study procedures, and voluntary provision of written informed consent.

Exclusion Criteria:

* Patients will be excluded if they meet any of the following conditions: inability to cooperate with awake intubation due to severe anxiety, cognitive impairment, or psychiatric disorders; a history of total laryngectomy or loss of normal laryngeal anatomical structures that precludes oral or nasal flexible bronchoscopic intubation; severe coagulation disorders or an uncontrollable risk of bleeding; or any other condition deemed by the investigators to make participation inappropriate, such as refusal of video recording or special confidentiality requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with laryngeal cancer or laryngeal tumors scheduled for laryngeal surgery under general anesthesia, who are assessed preoperatively as requiring awake flexible bronchoscopic intubation for airway safety. All participants will undergo routine clinical management without alteration of anesthetic strategy, with additional standardized video recording during awake intubation for observational analysis.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
proportion of cases | During the awake flexible bronchoscopic intubation procedure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. McTigue C, McGoldrick KE，Airway management in head and neck cancer: A review. Curr Opin Anaesthesiol. 2021;34(1):41-49. 2. Awake fiberoptic intubation in the management of the difficult airway. Anesth Analg. 2001;92(6):1523-1528. 3. Awake tracheal intubation: a modern, high-value technique in airway management.Br J Anaesth. 2023;130(2):e151-e154. 4. Cook TM, Woodall N, Frerk C, et al. Major complications of airway management in the United Kingdom: results of the 4th National Audit Project (NAP4). Br J Anaesth. 2011;106(5):617-631. 5. Ozgul G, Cetinkaya E, Ozgul MA, et al. Efficacy and safety of electromagnetic navigation bronchoscopy with or without radial endobronchial ultrasound for peripheral lung lesions. Endosc Ultrasound. 2016;5:189-195. 6. Ahmad I, El-Boghdadly K, Bhagrath R, et al. Difficult Airway Society guidelines for awake tracheal intubation (ATI) in adults. Anaesthesia. 2020;75(4):509-528. 7. Rosenstock CV, Thøgersen B, Afshari A, Christensen AL, Eriksen C, Gätke MR. Awake fiberoptic or awake video laryngoscopic tracheal intubation in patients with anticipated difficult airway management: a randomized clinical trial. Anesthesiology. 2012;116(6):1210-1216. 8. Kramer A, Muller D, Pfannenstiel C, Mohr C, Groeben H. Fibreoptic vs videolaryngoscopic (C-MAC D-BLADE) nasal awake intubation in head and neck cancer patients with difficult airways - a randomized clinical trial.Anaesthesia. 2015;70(12):1311-1316. 9. Mendonca C, Mesbah A, Velayudhan A, Danha R. A randomized clinical trial comparing the flexible fibrescope and the Pentax Airway Scope® for awake oral tracheal intubation. Anaesthesia. 2016;71(8):908-914.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT07324317/Prot_SAP_000.pdf